CLINICAL TRIAL: NCT04059341
Title: Early Extracorporeal Shockwave Therapy for Erectile Dysfunction in Radically Prostatectomised Men.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lund,MD, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ELIESWTEDRP
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Erectile Dysfunction; Extracorporeal Shockwave Therapy; Radical Prostatectomy
Keywords: Radical Prostatectomy; Prostatectomy; Nerve-sparing; Non nerve-sparing; Erectile dysfunction; Erectile function; Shockwave; LI-ESWT; ESWT; Low intensity extracorporeal shockwave therapy; extracorporeal shockwave therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomised, single-blinded, placebo-controlled trial
Who Masked: Participant
Masking Description: Sham LI-ESWT treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active LI-ESWT (Experimental): Active group receives five sessions of low intensity extracorporeal shockwave treatment, once per week for five consecutive weeks. Treatment is initiated three weeks after radical prostatectomy and is given using DUOLITH® SD1 manufactured by STORZ MEDICAL AG.
  Interventions: Device: Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT)
- Sham (Sham Comparator): Sham group receives five sessions of sham low intensity extracorporeal shockwave treatment, once per week for five consecutive weeks. Treatment is initiated three weeks after radical prostatectomy and is given using DUOLITH® SD1 manufactured by STORZ MEDICAL AG with a shockwave absorbing adapter.
  Interventions: Device: Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT)

INTERVENTIONS:
Device: Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT) — Five sessions of penile Low Intensity Extracorporeal Shockwave Therapy initiated three weeks after radical prostatectomy.

SUMMARY:
The purpose of this project is to assess the relationship between low intensity shock wave treatment (LI-SWT) and erectile function (ED) in patients who have undergone radical prostatectomy (RP).

ELIGIBILITY:
Inclusion Criteria:

* Radically prostatectomised men
* Non nerve-sparing or nerve-sparing RP.
* Age 20-80 years
* Have been in a relationship for more than 3 months.
* Sexually active
* Patient can give informed consent.

Exclusion Criteria:

* Men with ED of neuropathological or psychogenic origin
* Rectal extirpation, radiation therapy to the pelvic area and recovery from any other cancer within the past 5 years are excluded.
* Patients with heart disease prohibiting sexual activity or taking medication with antiandrogens, anticoagulant (apart from aspirin) or systemic use of glucocorticoids within 5 weeks.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 Score 1 | One month after final treatment session
  Change in International Index of Erectile Function (IIEF-5) score compared to baseline
IIEF-5 Score 3 | Three months after final treatment session
  Change in International Index of Erectile Function (IIEF-5) score compared to baseline
IIEF-5 Score 6 | Six months after final treatment session
  Change in International Index of Erectile Function (IIEF-5) score compared to baseline

SECONDARY OUTCOMES:
EDITS | One month after final treatment session
  Erectile Dysfunction Inventory of Treatment Satisfaction score
RigiScan | One month after final treatment session
  Change in nocturnal erections compared to baseline
EHS 1 | One month after final treatment session
  Change in Erection Hardness Score compared to baseline
EHS 3 | Three months after final treatment session
  Change in Erection Hardness Score compared to baseline
EHS 6 | Six months after final treatment session
  Change in Erection Hardness Score compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No